CLINICAL TRIAL: NCT07336134
Title: Uptake of HPV Self-sampling in Underserved Minority Women Using a Community Health Worker Model: Comparison of Evalyn Brush and Copan Floqswab
Brief Title: PopSci CHW4CervixHealth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: iRISID-2025-0275; JT 44840 (Other: JeffTrial Number)
Record Dates: First submitted 2025-11-07; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Cervical Cancer; Hpv; Human Papilloma Virus; HPV Infection
Keywords: Copan FLOQswab; Evalyn® Brush; HPV self-collection; self-collection; community health workers; underscreened women; concordance
MeSH Terms: conditions — Uterine Cervical Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Intervention Model Description: Phase I: The validation consists of patients using a self-sample kit at their scheduled Pap smear at Jefferson OBGYN.
  Phase II: The CHW4CervixHealth intervention consists of CHW facilitated culturally-tailored community workshops about cervical health and cervical cancer prevention, distribution and collection of HPV self-collection, and follow-up from results when appropriate.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Arm 1: Evalyn Brush Self-Collection - Phase I (Validation) (Experimental): Participants will be provided the Evalyn Brush self-sample kit at their scheduled Pap smear; a self-collected HPV test will also be collected as part of validation purposes for the study. Results will be shared from both their regularly scheduled appointment and the HPV self sample kit.
  Interventions: Device: Evalyn® Brush
- Arm 2: Evalyn Brush Self-Collection - Phase II (Community Implementation) (Experimental): Participants will be assigned to use the Evalyn Brush device to evaluate feasibility and acceptability of use. Trained bilingual community health workers (CHWs) will provide culturally-tailored community workshops about cervical health and cervical cancer prevention, distribution and collection of HPV self-collection, and follow-up from results when appropriate.
  Interventions: Device: Evalyn® Brush; Behavioral: CHW4CervicalHealth
- Arm 3: Copan FLOQSwab Self-Collection - Phase II (Community Implementation) (Experimental): Participants will be assigned to use the Copan FLOQSwab device to evaluate feasibility and acceptability of use. Trained bilingual community health workers (CHWs) will provide culturally-tailored community workshops about cervical health and cervical cancer prevention, distribution and collection of HPV self-collection, and follow-up from results when appropriate.
  Interventions: Device: Copan Floqswab; Behavioral: CHW4CervicalHealth

INTERVENTIONS:
Device: Evalyn® Brush — Participants use Evalyn® Brush device to collect a cervical sample for HPV testing.
  Other Names: Rovers® Self-Sampling Device; simply Evalyn; Viba-Brush®
  Arms: Arm 1: Evalyn Brush Self-Collection - Phase I (Validation); Arm 2: Evalyn Brush Self-Collection - Phase II (Community Implementation)
Device: Copan Floqswab — Participants use the Copan Floqswab device to collect a cervical sample for HPV testing.
  Other Names: 4N6FLOQSwabs® Genetics; eSwab®; hDNA Free FLOQSwabs®; flocked swabs; nylon-tipped swabs
  Arms: Arm 3: Copan FLOQSwab Self-Collection - Phase II (Community Implementation)
Behavioral: CHW4CervicalHealth — The CHW4CervicalHealth intervention is a community health care worker (CHW)-led education and support program designed to promote HPV self-collection among underserved women. Trained bilingual CHWs provide culturally-tailored community workshops about cervical health and cervical cancer prevention, distribution and collection of HPV self-collection, and follow-up from results when appropriate.
  Arms: Arm 2: Evalyn Brush Self-Collection - Phase II (Community Implementation); Arm 3: Copan FLOQSwab Self-Collection - Phase II (Community Implementation)

SUMMARY:
Phase I: Validating self-collection kit by comparing their results with clinical Pap smear results in a cohort of 20 patients.

Phase II: Evaluate the feasibility and acceptability of the CHW4CervicalHealth: Use of a self-collection kit to improve cervical health screening intervention aimed to promote HPV self-collection uptake among screening-eligible and under-screened ethnic minority women in the community.

DETAILED DESCRIPTION:
The self-collection kits will be collected at the clinic (Phase I) or at the end of the workshop (Phase II). A chain-of-custody form for each kit will be associated with the specimen and the clinic nurse will label and prepare to transport them via courier to the Jefferson NJ Molecular Virology lab, Cherry Hill, NJ; Richard Sunday, Lab Supervisor, will process according to Roche, the self-collected vaginal specimens suspended in PreservCyt® may be stored at 2-30°C (35.6- 86°F) for up to 1 month after the date of collection.

Phase I: In person accrual, enrollment and study implementation will take 15-30 minutes.

-Clinic staff will collect self-collection kit at appointment.

Phase II: Workshops will take about 30 minutes to complete and another 30 minutes to complete survey and self-collection kit use.

* Conduct educational workshops in participants primary language
* For those choosing to use the self-sample kit, obtain and document e-consent or paper consent from potential participants in their primary language.
* Provide participants with self-collection testing kits during workshop along with instructions
* Collect self-collection kit samples from participants and place in pre-made sample bags with appropriate label. CHW will take custody and coordinate with OBGYN clinic staff to drop off self-collected samples
* Collect post workshop survey and conduct post workshop interviews or focus group
* OBGYN staff set-up courier to send samples to NJ lab

ELIGIBILITY:
Inclusion Criteria:

Phase I:

* Women aged 25-65 years
* Scheduled for a Pap smear test appointment at Jefferson OBGYN Center City location
* Willing and able to provide informed consent for participation in the study
* Agree to perform an HPV self-collection collection procedure during the same visit
* Have not undergone a hysterectomy (intact cervix required)

Phase II:

This intervention targets under-screened minority individuals who must meet all the following inclusion criteria to be eligible to participate in the study:

* Women aged 25-65 years
* Who has not had a Pap smear in the past three to five years based on age of prior screening and type of screening. If under the age of 30, in the past 3 years and if over the age of 30, in the past 5 years. Participant will self-report normal pap smear and date.
* Self-identify as Hispanic, Black/African or Black Caribbean, Chinese, Korean, or Vietnamese
* Competent to give consent and provide signed and dated informed consent form in their preferred language.

Exclusion Criteria:

Phase I:

* Current pregnancy (self-reported or confirmed)
* Previous participation in an HPV self-collection study within the past 12 months
* Presence of visible vaginal or cervical infection or symptoms suggestive of a current genital tract infection
* Inability to comply with study procedures or follow instructions (e.g., due to language barriers or cognitive impairments)

Phase II:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Have a history of hysterectomy, cervical cancer
* Self-report participation in a cervical cancer screening or other prevention study
* Pregnant (self-reported)
* Inability to provide informed consent

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Concordance of Self-Collected vs. Clinically collected sample (Phase I) | at the visit (approximately 30 minutes) and analysis completed within 2 weeks
  Concordance rate between self-collection kit results and clinical Pap smear findings (measured as agreement in detection of HPV and/or abnormal cytology). Agreement between the two methods will be evaluated using Cohen's kappa statistic, with values interpreted based on standard benchmarks for strength of agreement. Sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) will be calculated to determine the accuracy of self-collection kits relative to the clinician-collected gold standard.
Feasibility of HPV Self-Collection: Completion of Self-Collection Kit | Within 12 months
  Feasibility will be assessed as the number of participants who proceed with HPV self-collection using the study kit out of the total number of participants enrolled in the study.

SECONDARY OUTCOMES:
Change in Participants' HPV-related knowledge and perceived comfort with self-collection | From Baseline to Post-Intervention (approximately 18 months)
  Paired sample t-tests will analyze changes in knowledge scores from baseline to post-intervention. Statistical analysis will be conducted using SPSS 25, with significance set at p < .05.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Dayaratna, MD, MBA, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States